CLINICAL TRIAL: NCT03482947
Title: TAP vs Caudal Block Using Dexmedetomidine/Bupivacaine Combination for Postoperative Analgesia in Pediatric Patients Undergoing Unilateral Inguinal Hernia Repair
Brief Title: TAP vs Caudal Block Using Dexmedetomidine/ Bupivacaine for Post Operative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, MD, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TAP/ECB
Record Dates: First submitted 2018-03-18; First posted 2018-03-29 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Analgesia, Epidural
Keywords: Dexmedetomidine; pediatrics; postoperative;; Analgesia; caudal
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP (Experimental): ultrasonography-guided transversus abdominis plane block administration of (1 mL/kg of bupivacaine 0.25% plus 1 μ/kg dexmedetomidine).
  Interventions: Drug: ultrasonography-guided TAP block
- Caudal (Experimental): Caudal epidural block administration of (1 mL/kg of bupivacaine 0.25% &1 μ/kg dexmedetomidine
  Interventions: Drug: Caudal epidural block

INTERVENTIONS:
Drug: ultrasonography-guided TAP block — (1 mL/kg of bupivacaine 0.25% plus 1 μ/kg dexmedetomidine).
  Arms: TAP
Drug: Caudal epidural block — (1 mL/kg of bupivacaine 0.25% plus 1 μ/kg dexmedetomidine)
  Arms: Caudal

SUMMARY:
Caudal epidural block is a well-established and commonly performed regional neuraxial technique for providing intraoperative and postoperative analgesia in children scheduled for lower abdomen/perineal surgical interventions. Although the efficacy and safety of Caudal epidural block are fairly high, the associated complications, such as inadvertent dural puncture, unwarranted motor blockade of the lower limbs, and disturbance of bladder function, limit its use. Furthermore, a major limitation of an uncomplicated Caudal epidural block when administered as a "single-shot" technique is its brief duration of action (up to 6 hours), which makes administration of additional analgesics necessary .

DETAILED DESCRIPTION:
Ultrasonography guidance, by virtue of real-time visualization of the muscle layers and fascial planes, has significantly facilitated practice of regional nerve blockade for it offers confirmation of the spread of the local anesthetic drug in the correct space. Interestingly, there has been a reinvigoration of interest in ultrasonography-guided transversus abdominis plane block in children since its emergence as a valid postoperative analgesia alternative in adults undergoing abdominal surgery. transversus abdominis plane block involves blockade of spinal afferent nerves in the neurofascial plane between the internal oblique and transversus abdominis muscle. Whereas the advantages (reduction in pain intensity/analgesic requirements) of ultrasonography-guided transversus abdominis plane block have been well documented in adults in the first 48 hours post surgery, in children, its use as a primary postoperative analgesia technique remains limited. Caudal anesthesia is easy to perform in younger children; however, its main disadvantage is the short duration of action. Even bupivacaine, along-acting local anesthetic drug, can provide only4-8 h of analgesia. Dexmedetomidine is a highly selective alfa2 agonist with sedative and analgesic properties. It has an alfa1/2 selectivity ratio of 1600 : 1, which is eight times more potent than clonidine (200 : 1)[16]. DEX has been used effectively in intensive care to aid weaning from mechanical ventilation and is being used increasingly in children

ELIGIBILITY:
Inclusion Criteria:

* patients 2-8 years

Exclusion Criteria:

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia. | 24 hours
  time for first analgesic request

SECONDARY OUTCOMES:
Postoperative analgesia | 24 hours
  total amount analgesic administered
Postoperative pain | 24 hours
  using the FLACC scale.Rate child on each of the five categories (face, legs, arms, crying, consolability). Each category is scored on the 0 to 2 scale. Add the scores together (for a total possible score of 0 to 10).

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

REFERENCES:
- [Result] Tsui BC, Berde CB. Caudal analgesia and anesthesia techniques in children. Curr Opin Anaesthesiol. 2005 Jun;18(3):283-8. doi: 10.1097/01.aco.0000169236.91185.5b. PMID 16534352
- [Result] Koul A, Pant D, Sood J. Caudal clonidine in day-care paediatric surgery. Indian J Anaesth. 2009 Aug;53(4):450-4. PMID 20640207
- [Result] Suresh S, Long J, Birmingham PK, De Oliveira GS Jr. Are caudal blocks for pain control safe in children? an analysis of 18,650 caudal blocks from the Pediatric Regional Anesthesia Network (PRAN) database. Anesth Analg. 2015 Jan;120(1):151-156. doi: 10.1213/ANE.0000000000000446. PMID 25393589
- [Result] Menzies R, Congreve K, Herodes V, Berg S, Mason DG. A survey of pediatric caudal extradural anesthesia practice. Paediatr Anaesth. 2009 Sep;19(9):829-36. doi: 10.1111/j.1460-9592.2009.03116.x. PMID 19691690